CLINICAL TRIAL: NCT05805917
Title: Comparative Clinical Trial on Neoviderm Skin Emulsion and Connettivina 0.2% Cream to Evaluate the Normalization Process of the Skin and Reduction of Cutaneous Tension and Pain in Patients With Superficial Burns Grade 1 and 2
Brief Title: Comparative Clinical Trial on Neoviderm Skin Emulsion and Connettivi-na 0.2% Cream to Evaluate the Normalization Process of the Skin and Re-duction of Cutaneous Tension and Pain in Patients With Superficial Burns Grade 1 and 2
Acronym: NVD01/22
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istituto Ganassini S.p.A. di Ricerche Biochimiche (Industry)
Responsible Party: Sponsor
Organization: Ganassini Corporate (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NVD01/22
Record Dates: First submitted 2023-03-21; First posted 2023-04-10 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Dermatology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 25 subjects treated with Neoviderm Skin Emulsion (Experimental)
  Interventions: Device: Neoviderm Skin Emulsion medical device
- 25 patients treated with Connettivina 0.2% Cream (Active Comparator)
  Interventions: Drug: Connettivina 0.2% Cream

INTERVENTIONS:
Device: Neoviderm Skin Emulsion medical device — Neoviderm Skin Emulsion will be applied twice daily, to cover the entire cutaneous surface interested by burns, followed by a gentle massage to spread the product evenly of all the affected skin.
  Arms: 25 subjects treated with Neoviderm Skin Emulsion
Drug: Connettivina 0.2% Cream — Connettivina 0.2% Cream will be applied twice daily, to cover the entire cutaneous surface interested by burns, followed by a gentle massage to spread the product evenly of all the affected skin.
  Arms: 25 patients treated with Connettivina 0.2% Cream

SUMMARY:
It is a single centre, randomized (set up or distributed in a deliberately random way), open-label (study participants and researchers both know which treatment the patient is receiving), prospective, interventional, post-marketing, controlled (An experiment or clinical trial in which two groups are used for comparison purpose), non-inferiority study (a study that tests whether a new treatment is not worse than an active treatment it is being compared to).

The PRIMARY OBJECTIVE is to assess the reduction of skin tension in patients with 1st and 2nd degree superficial burns treated either with Neoviderm Skin Emulsion medical device or Connettivina 0.2% Cream.

Neoviderm Skin Emulsion soothes and relieves the skin, promoting its physiological normalization process. It is suitable for adults, children and infants in case of sunburns; 1st degree and 2nd degree superficial burns; superficial ulcers; protection before and after radiotherapy treatment; skin irritation and manifestations involving redness; skin cracks, including recurring ones; desquamative states; erythema; dry skin; small abrasions. It is also indicated only for adults in case of tattoo aftercare and chemical peel.

DETAILED DESCRIPTION:
Investigation Title:

Comparative clinical trial on Neoviderm Skin Emulsion and Connettivina 0.2% Cream to evaluate the normalization process of the skin and reduction of cutaneous tension and pain in patients with superficial burns grade 1 and 2.

Sponsor:

Istituto Ganassini S.p.A.di Ricerche Biochimiche

Medical Device:

Neoviderm Skin Emulsion - Medical Device class IIb

Intended Use:

Because of its protective and moisturizing action, Neoviderm Skin Emulsion soothes and relieves the skin, promoting its physiological normalization process. It is suitable for adults, children and infants in case of sunburns; 1st degree and 2nd degree superficial burns; superficial ulcers; protection before and after radiotherapy treatment; skin irritation and manifestations involving redness; skin cracks, including recurring ones; desquamative states; erythema; dry skin; small abrasions. It is also indicated only for adults in case of tattoo aftercare and chemical peel.

Background and Rationale:

First degree burns (sometimes also called "superficial" burns) are usually limted to the epidermis, while partial thickness burns (also called 2nd degree burns) involve part of the dermis and can be superficial or deep.

Partial thickness burns involve the papillary dermis (the most superficial portion). These burns heal in 1-2 weeks and the scar is usually minimal. The healing process starts from the cells of the epidermis that line the ducts of the sweat glands and the hair follicles; these cells grow from the surface, migrate along the surface to meet cells from nearby glands and follicles.

Superficial first- and second-degree burns are therefore attributable to minor or minor burns. The severity of the burn also depends on its extent: localized burns are those in which the body surface involved is ≤ 20% in adults, ≤15% in children 10-15 years of age, ≤10 % in children 3-10 years of age and seniors over 65 years of age.

Scientific evidence therefore supports the rationale for developing a medical device (Neoviderm Skin Emulsion) aimed at restoring the integrity of the injured skin by reducing tension and pain, characteristic manifestations of first degree and second-degree superficial burns. Therefore, the study is aimed to evaluate the comparative activity of the Neoviderm Skin Emulsion, Medical Device class IIb and Connettivina 0.2% Cream, OTC product.

Overall Study Design:

It is a single centre, randomized, open-label, prospective, interventional, post-marketing, controlled, non-inferiority study.

PRIMARY OBJECTIVE:

to assess the reduction of skin tension in patients with 1st and 2nd degree superficial burns treated either with Neoviderm Skin Emulsion medical device or Connettivina 0.2% Cream.

SECONDARY OBJECTIVE:

to assess the reduction of pain sensation in patients with 1st and 2nd degree superficial burns treated either with Neoviderm Skin Emulsion medical device or Connettivina 0.2% Cream.

EXPLORATORY OBJECTIVE:

to assess the health status of skin in patients with 1st and 2nd degree superficial burns treated either with Neoviderm Skin Emulsion medical device or Connettivina 0.2% Cream.

Primary Endpoint:

To compare the reduction in skin tension by means of a corneometer, at baseline (V0) and after 14 days of treatment (V2), in patients with 1st and 2nd degree superficial burns treated either with Neoviderm Skin Emulsion medical device or Connettivina 0.2% Cream.

Secondary Endpoint:

To compare the reduction in pain by means of a Visual Analogue Scale (VAS), at baseline (V0) and after 14 days of treatment (V2), in patients with 1st and 2nd degree superficial burns treated either with Neoviderm Skin Emulsion medical device or Connettivina 0.2% Cream.

Exploratory Endpoint:

To assess the health status of the skin, by analysing images obtained through videodermatoscopy at the baseline (V0) and after 14 days of treatment (V2), in patients with 1st and 2nd degree superficial burns treated either with Neoviderm Skin Emulsion medical device or Connettivina 0.2% Cream.

Sample size:

50 subjects (25 subjects treated with Neoviderm Skin Emulsion and 25 patients treated with Connettivina 0.2% Cream).

Dosing:

The two products (Neoviderm Skin Emulsion and Connettivina 0.2% Cream) will be applied twice daily, to cover the entire cutaneous surface interested by burns, followed by a gentle massage to spread the product evenly of all the affected skin.

Statistical Consideration

Decriptive statistics will be summarized, for entire population and separately per treatment groups, according to the type of variable:

* for quantitative variables: standard quantitative statistics (N, mean, standard deviation, median, interquartile range, minimum and maximum);
* for qualitative variables: frequency distribution [number of non-missing observations (N) and percentages (%)].

For inferential tests of the difference between groups:

* for quantitative variables (difference of two means or medians): unpaired T-tests (or the corresponding non-parametric Wilcoxon-Mann-Whitney tests, as appropriate) will be performed;
* for qualitative variables (difference of proportions): Chi-Square tests or Fisher's exact tests will be performed.

The number of adverse events (AEs) and the number and proportion of patients with at least one AE will be presented, both for entire population and separately per groups.

ELIGIBILITY:
Inclusion Criteria:

The patients should comply with all the following inclusion criteria.

* Adult subjects, adolescents between 11 and 17 years, and children aged ≥ 3 years.
* Both sexes (males and females).
* Subjects or subjects'parents that have given the appropriate writ-ten informed consent (in accordance with local requirements) for the participation in the study at the time of enrolment,
* Subjects with 1st and 2nd superficial burns, either of physical or liquid burns, with an affected cutaneous area ≤ 20% in adults, ≤ 15% in children between 10 and 15 years of age, and ≤ 10% in children between 3 and 10 years and seniors over 65 years of age.

Exclusion Criteria:

Patients with any one of the following exclusion criteria are not eligible:

* Subjects with chemically induced burns.
* Subjects with electrically induced burns.
* Hypersensitivity to the active ingredients of products under study, or to one or more excipients present in the products under study or known hypersensitivity to any other product containing the same active ingredients or excipients.
* Subjects with concomitant infection of the affected burn or in-fected lesions and / or bleeding.
* General disorders that can affect the safety or well-being of the subject or interfere with the response of the skin.
* Current participation in another trial is not permitted unless it is a non-interventional study, and the sole purpose of the trial is for long-term follow up describing clinical features or survival data (registry).
* Women who are known to be pregnant or breastfeeding.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-04-17 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
To compare the change in skin tension by means of a corneometer, at baseline (V0) and after 14 days of treatment (V2). Change will be assessed | At Screening (V0 Randomization and treatment will be assigned) and at V2 (day 14 after treatment). Change will be assessed
  To compare the change in skin tension by means of a corneometer, at baseline (V0) and after 14 days of treatment (V2), in patients with 1st and 2nd degree superficial burns treated either with Neoviderm Skin Emulsion medical device or Connettivina 0.2% Cream. Change will be assessed

SECONDARY OUTCOMES:
To compare the change in pain by means of a Visual Analogue Scale (VAS), at baseline (V0) and after 14 days of treatment (V2). Changed will be assessed. | At Screening (V0 Randomization and treatment will be assigned) and at V2 (day 14 after treatment). Change will be assessed
  To compare the change in pain by means of a Visual Analogue Scale (VAS), at baseline (V0) and after 14 days of treatment (V2), in patients with 1st and 2nd degree superficial burns treated either with Neoviderm Skin Emulsion medical device or Connettivina 0.2% Cream.
To assess the health status of the skin. The measurement tool will be videodermatoscopy that will notice morphological qualities diagnosing skin changes at the baseline (V0) and after 14 days of treatment (V2). Changed will be assessed. | At Screening (V0 Randomization and treatment will be assigned) and at V2 (day 14 after treatment). Change will be assessed
  To assess the health status of the skin. The measurement tool will be videodermatoscopy that will notice morphological qualities diagnosing skin changes at the baseline (V0) and after 14 days of treatment (V2). Currently, videodermatoscopy is the most advanced, non invasive method of diagnosing skin changes. It involves displaying the area being studied, most often a nevus, on a computer screen magnified up to 200 times, thus making it possible to notice its morphological qualities not visible to the human eye.
  Patients with 1st and 2nd degree superficial burns will be treated either with Neoviderm Skin Emulsion medical device or Connettivina 0.2% Cream.

CONTACTS AND LOCATIONS:
Locations (1):
- UO Dermatologia - Piraccini IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Undecided